CLINICAL TRIAL: NCT02576990
Title: A Phase II Study of Pembrolizumab (MK-3475) in Subjects With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) or Relapsed or Refractory Richter Syndrome (rrRS)
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma or Relapsed or Refractory Richter Syndrome (MK-3475-170/KEYNOTE-170)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-170; MK-3475-170 (Other: Merck); KEYNOTE-170 (Other: Merck); 2015-002406-37 (EudraCT Number)
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Mediastinal Large B-cell Lymphoma; Richter Syndrome
Keywords: Programmed Cell Death 1 (PD-1, PD1); Programmed Cell Death-Ligand 1 (PD-L1, PDL1); Programmed Cell Death-Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (Experimental): Participants with rrPMBCL receive pembrolizumab 200 mg every 3 weeks (Q3W), intravenous infusion (IV) on Day 1 of each 3-week cycle for up to a maximum of 35 administrations (approximately 2 years).
  Interventions: Biological: Pembrolizumab
- Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS) (Experimental): Participants with rrRS receive pembrolizumab 200 mg Q3W, IV for each 3-week cycle for up to a maximum of 35 administrations (approximately 2 years). Effective with Protocol Amendment 04, enrollment into this cohort was closed.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®; SCH 900475

SUMMARY:
In this study, participants with relapsed or refractory primary mediastinal large B-cell lymphoma (rrPMBCL) or relapsed or refractory Richter Syndrome (rrRS) will receive pembrolizumab (MK-3475). The efficacy of pembrolizumab in the treatment of rrPMBCL and rrRS will be evaluated. The primary study hypothesis is that intravenous (IV) administration of single agent pembrolizumab to the rrPMBCL cohort will result in an Objective Response Rate (ORR) of greater than 15% using the International Working Group (IWG) response criteria (Cheson, 2007) by independent central review.

Effective with Protocol Amendment 04, enrollment into the rrRS cohort was closed.

DETAILED DESCRIPTION:
Treatment with pembrolizumab will continue for a maximum of 35 administrations (approximately 2 years) or until documented disease progression by investigator assessment, unacceptable adverse event(s) (AEs), intercurrent illness that prevents further administration of treatment, participant withdraws consent, pregnancy of the participant, noncompliance with study treatment or procedure requirements, or administrative reasons.

ELIGIBILITY:
Inclusion Criteria:

* Primary mediastinal large B-cell lymphoma (PMBCL):
* Diagnosis of relapsed or refractory primary mediastinal large B-cell lymphoma (rrPMBCL) AND
* Has relapsed after autologous stem cell transplant (auto-SCT) or has failed to achieve a Complete Response or Partial Response within 60 days of auto-SCT. Participants may have received intervening therapy after auto-SCT for relapsed or refractory disease, in which case they must have relapsed after or be refractory to their last treatment OR
* For participants who are ineligible for auto-SCT, has received at least ≥2 lines of prior therapy and has failed to respond to or relapsed after their last line of treatment. For participants who received consolidative local radiotherapy after systemic therapy, local radiotherapy will not be considered as a separate line of treatment
* Previously exposed to rituximab as part of prior lines of treatment
* Richter syndrome (RS):
* Pathologic diagnosis per local institutional review of RS that transformed from chronic lymphocytic leukemia (CLL)
* Relapsed or refractory Richter syndrome and has received ≥1 previous treatment for RS
* All Participants:
* Radiographically measurable disease
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Life expectancy >3 months
* Adequate organ function
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug
* Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug
* Is receiving systemic steroid therapy <3 days before the first dose of study drug or receiving any other form of immunosuppressive medication
* Prior monoclonal antibody within 4 weeks prior to study Day 1 (2 weeks for RS participants) or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier (2 weeks for RS participants)
* Prior chemotherapy or targeted small molecule therapy within 2 weeks prior to study Day 1 or prior radiation therapy within 4 weeks prior to study Day 1
* Allogeneic hematopoietic stem cell transplantation within the last 5 years.
* Has a known additional malignancy (except underlying CLL for RS) that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Known clinically active central nervous system involvement
* Active autoimmune disease requiring systemic treatment in past 2 years
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis
* Active infection requiring intravenous systemic therapy
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study drug
* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), anti-programmed cell death ligand 2 (anti-PD-L2), anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Known human immunodeficiency virus (HIV), or Hepatitis B or C
* Has received a live vaccine within 30 days prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Armand P, Rodig S, Melnichenko V, Thieblemont C, Bouabdallah K, Tumyan G, Ozcan M, Portino S, Fogliatto L, Caballero MD, Walewski J, Gulbas Z, Ribrag V, Christian B, Perini GF, Salles G, Svoboda J, Zain J, Patel S, Chen PH, Ligon AH, Ouyang J, Neuberg D, Redd R, Chatterjee A, Balakumaran A, Orlowski R, Shipp M, Zinzani PL. Pembrolizumab in Relapsed or Refractory Primary Mediastinal Large B-Cell Lymphoma. J Clin Oncol. 2019 Dec 1;37(34):3291-3299. doi: 10.1200/JCO.19.01389. Epub 2019 Oct 14. PMID 31609651
- [Result] Armand P, Murawski N, Molin D, Zain J, Eichhorst B, Gulbas Z, Hawkes EA, Pagel JM, Phillips T, Ribrag V, Svoboda J, Stathis A, Chatterjee A, Orlowski R, Marinello P, Christian B. Pembrolizumab in relapsed or refractory Richter syndrome. Br J Haematol. 2020 Jul;190(2):e117-e120. doi: 10.1111/bjh.16762. Epub 2020 Jun 16. No abstract available. PMID 32544980
- [Result] Zinzani PL, Thieblemont C, Melnichenko V, Bouabdallah K, Walewski J, Majlis A, Fogliatto L, Garcia-Sancho AM, Christian B, Gulbas Z, Ozcan M, Perini GF, Ghesquieres H, Shipp MA, Thompson S, Chakraborty S, Marinello P, Armand P. Pembrolizumab in relapsed or refractory primary mediastinal large B-cell lymphoma: final analysis of KEYNOTE-170. Blood. 2023 Jul 13;142(2):141-145. doi: 10.1182/blood.2022019340. PMID 37130017
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 80 participants allocated in the study, 76 participants received at least one dose of study treatment.
Groups:
- Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL): Pembrolizumab 200 mg every 3 weeks (Q3W), intravenous infusion (IV) on Day 1 of each 3-week cycle for up to 35 administrations (approximately 2 years).
- Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS): Pembrolizumab 200 mg Q3W, IV on Day 1 of each 3-week cycle for up to 35 administrations (approximately 2 years).
Period: Overall Study
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Started | 56 | 24
Treated | 53 | 23
Completed | 0 | 0
Not Completed | 56 | 24
Not completed — Death | 29 | 18
Not completed — Physician Decision | 1 | 0
Not completed — Screen failure | 2 | 0
Not completed — Sponsor's decision | 24 | 4
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All allocated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS) | Total
Number analyzed (Participants) | 56 | 24 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.0 (10.4) | 67.2 (11.0) | 44.7 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 7 | 37
  Male | 26 | 17 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 37 | 21 | 58
  Unknown or Not Reported | 15 | 2 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 51 | 24 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on International Working Group (IWG) Response Assessment Criteria Per Independent Central Review
Description: The ORR was assessed by independent central review utilizing the International Working Group [IWG] response assessment criteria per Cheson 2007 of pembrolizumab in participants with rrPMBCL. For participants with rrRS, IWG criteria with special considerations for RS was used for progression. The ORR was defined as the percentage of participants who had a response (complete response, CR or partial response, PR) prior to disease progression. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. Participants with missing data were considered non-responders. In the rrPMBCL cohort, an exact binomial test was conducted versus a fixed historical control rate. For the rrPMBCL cohort, the ORR was estimated as well as a 95% 2-sided exact confidence interval (CI) using the Clopper-Pearson method whereas the rrRS cohort was estimated with a 90% 2-sided CI.
Time Frame: Up to approximately 27 months (Database Cutoff: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Percentage of participants | 45.3 [31.6 to 59.6] | 13.0 [3.7 to 30.4]

2. Secondary Outcome: ORR Based on IWG Response Assessment Criteria by Investigator Assessment
Description: The ORR was assessed by Investigator assessment utilizing the IWG response assessment criteria per Cheson 2007 of pembrolizumab in participants with rrPMBCL. For participants with rrRS, IWG criteria with special considerations for RS was used for progression. The ORR was defined as the percentage of participants who had a response (CR or PR) prior to disease progression. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. Participants with missing data were considered non-responders. In the rrPMBCL cohort, an exact binomial test was conducted versus a fixed historical control rate.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Percentage of participants | 41.5 [30.0 to 53.7] | 4.3 [0.2 to 19.0]

3. Secondary Outcome: Progression Free Survival (PFS) Based on IWG Response Assessment Criteria by Independent Central Review
Description: PFS was defined as the time from first dose to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PD is the appearance of any new lesion or increase by ≥ 50% of previously involved site from nadir. Calculated from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Months | 5.5 [2.8 to 15.1] | 1.6 [1.0 to 2.1]

4. Secondary Outcome: Progression Free Survival (PFS) Based on IWG Response Assessment Criteria by Investigator Assessment
Description: PFS was defined as the time from the first dose to the first documented PD or death due to any cause, whichever occurs first. PD is the appearance of any new lesion or increase by ≥ 50% of previously involved site from nadir. Calculated from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Months | 4.3 [2.8 to 13.8] | 1.8 [1.0 to 2.1]

5. Secondary Outcome: Duration of Response (DOR) Based on IWG Response Assessment Criteria by Independent Central Review in Participants With Responses
Description: The DOR was defined, only for the subgroup of participants who achieved a CR or PR by independent central review, as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of PD or to death due to any cause, whichever comes first. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. PD is the appearance any new lesion or increase by ≥ 50% of previously involved site from nadir. The analysis consisted of Kaplan-Meier estimates. DOR data was censored on the date of the last disease assessment documenting absence of PD for participants who did not have tumor progression and were still on study at the time of an analysis, were given antitumor treatment other than the study treatment, or were removed from study prior to documentation of tumor progression.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab) and who achieved a CR or PR by independent central review, as the time from start of the first documentation of objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 24 | 3
Months | NA [25.2 to NA] — NA = Median DOR was not reached (no progressive disease by time of last disease assessment). NA = DOR upper limit was not reached (no progressive disease by time of last disease assessment). | 4.5 [2.7 to 6.2]

6. Secondary Outcome: Duration of Response (DOR) Based on IWG Response Assessment Criteria by Investigator Assessment in Participants With Responses
Description: The DOR was defined, only for the subgroup of participants who achieved a CR or PR by investigator assessment, as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of PD or to death due to any cause, whichever comes first. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. PD is the appearance any new lesion or increase by ≥ 50% of previously involved site from nadir. The analysis consisted of Kaplan-Meier estimates. DOR data was censored on the date of the last disease assessment documenting absence of PD for participants who did not have tumor progression and were still on study at the time of an analysis, were given antitumor treatment other than the study treatment, or were removed from study prior to documentation of tumor progression.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab) and who achieved a CR or PR by investigator assessment, as the time from start of the first documentation of objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 24 | 1
Months | NA [25.2 to NA] — NA = Median DOR was not reached (no progressive disease by time of last disease assessment). NA = DOR upper limit was not reached (no progressive disease by time of last disease assessment). | NA [NA to NA] — NA = Median DOR was not reached (no progressive disease by time of last disease assessment). NA = DOR upper and lower limits were not reached (no progressive disease by time of last disease assessment).

7. Secondary Outcome: Disease Control Rate (DCR) Based on IWG Response Assessment Criteria by Independent Central Review
Description: The DCR was defined as the percentage of participants in the analysis population who have achieved a CR, PR or stable disease (SD) response prior to PD. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. SD is the failure to attain CR/PR or PD. PD is the appearance any new lesion or increase by ≥ 50% of previously involved site from nadir. Participants with missing data were considered non-responders.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Percentage of participants | 54.7 [42.6 to 66.5] | 17.4 [6.2 to 35.5]

8. Secondary Outcome: Disease Control Rate (DCR) Based on IWG Response Assessment Criteria by Investigator Assessment
Description: The DCR was defined as the percentage of participants in the analysis population who have achieved a CR, PR or SD response prior to PD. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites. SD is the failure to attain CR/PR or PD. PD is the appearance any new lesion or increase by ≥ 50% of previously involved site from nadir. Participants with missing data were considered non-responders.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Percentage of participants | 52.8 [40.7 to 64.7] | 26.1 [12.0 to 45.1]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose to death due to any cause. OS is presented from product limit (Kaplan-Meier) method for censored data (censored at the last assessment).
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Months | 22.3 [7.3 to NA] — NA = OS upper limit was not reached (insufficient number of deaths by time of last disease assessment). | 3.8 [1.8 to 18.1]

10. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who experienced an AE were reported.
Time Frame: Up to approximately 30 months (Up to 90 days after last dose of study treatment) (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Participants | 50 | 23

11. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who discontinued study drug due to an AE were reported.
Time Frame: Up to approximately 27 months (Database Cutoff Date: 28MAY2019)
Population: The analysis population included all participants who received at least one dose of study medication (pembrolizumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
Number analyzed (Participants) | 53 | 23
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs), non-serious AEs and all-cause mortality was collected up to approximately 56 months through end of trial (EOT) data cut-off date 23 Oct 2020.
Description: All-cause mortality was reported on all allocated participants. Serious and non-serious AEs were reported among participants who received at least one dose of study treatment. Per protocol, disease progression of cancer was not considered an AE unless related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to study drug were excluded.
Arm/Group | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS)
All-Cause Mortality (participants affected / at risk) | 30/56 | 19/24
Serious Adverse Events (participants affected / at risk) | 14/53 | 15/23
Other Adverse Events (participants affected / at risk) | 46/53 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (N=53) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS) (N=23)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab: Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (N=53) | Pembrolizumab: Relapsed or Refractory Richter Syndrome (rrRS) (N=23)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 7 (9)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 15 (29) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 3 (3)
Hypothyroidism (Endocrine disorders) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (8) | 6 (7)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Asthenia (General disorders) | 7 (10) | 2 (2)
Chest pain (General disorders) | 4 (4) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 6 (7) | 8 (8)
Pyrexia (General disorders) | 15 (25) | 3 (4)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (10) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 5 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 4 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 6 (11) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 2 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT02576990/Prot_SAP_001.pdf